CLINICAL TRIAL: NCT06540768
Title: Therapeutic Normothermia in the Treatment of Traumatic Brain Injury Trial: Feasibility Trial
Brief Title: Therapeutic Normothermia in TBI
Acronym: MAMBA-FT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre (Other)
Collaborators: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ian Ball, Dr., London Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14097
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Traumatic Brain Injury
Keywords: TBI; therapeutic normothermia; targeted temperature management; cognitive outcomes; traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Single center unblinded randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Therapeutic Normothermia Group (Active Comparator): Participants randomized to this group will be placed under a targeted temperature model aiming for normothermia for 72 hours. Temperature and interventions will be monitored every 4 hours for the entirety of the 24 hours. Participants will be followed post-discharge and will undergo cognitive assessments at 3 and 6 months.
  Interventions: Other: Therapeutic Normothermia Group
- Control Group (No Intervention): Participants randomized to this group will undergo usual care in the Critical Care Trauma Centre. Temperature will be monitored as per standard of care. Participants will be followed post-discharge and will undergo cognitive assessments at 3 and 6 months.

INTERVENTIONS:
Other: Therapeutic Normothermia Group — Maintenance of a body temperature between 35 and 37 degrees Celsius using conservative and pharmacological interventions for 72 hours.
  Arms: Therapeutic Normothermia Group

SUMMARY:
This feasibility trial is the first step in testing the hypothesis that maintenance of normal body temperature, called therapeutic normothermia (TN), for 72 continuous hours in traumatic brain injury (TBI) patients can improve cognitive function. The trial aims to answer the following questions:

1. Is it feasible to conduct this study? Conducting the trial includes the ability to identify and enroll appropriate participants, implement TN, and collect the required data.
2. Can the Creyos Health platform cognitive assessment tool be used to assess and quantify cognitive outcomes in TBI patients?

Researchers will address the aforementioned questions by looking at the following factors:

1. Identification and enrollment rates of appropriate patients
2. Implementation of the intervention and appropriate data collection while admitted
3. Accurate follow up and continued data collection post-discharge
4. Accessibility and ease of use of the Creyos Health platform cognitive assessment tool

Participants will undergo the following procedure:

1. Admission to the Critical Care Trauma Centre through the trauma service
2. Allocation to the intervention or no intervention group
3. Implementation of the intervention or of usual care for a continuous 72 hours
4. Completion of the Creyos Health platform cognitive assessment tool at 3 and 6 months post-discharge from the Critical Care Trauma Centre

DETAILED DESCRIPTION:
Therapeutic normothermia (TN) is globally accepted as standard of care in post-cardiac arrest patients to maximize neurologic recovery. Both hypothermia and normothermia have been trialed and were noted to prevent the harmful effects of hyperthermia on intracranial pressures and the cardiovascular system. Normothermia is favored for its improved cardiovascular, hematological, immunological, and metabolic outcomes. In trauma patients specifically, hypothermia (whether therapeutic or accidental) has been shown to result in worse outcomes and increased mortality. Despite this, therapeutic normothermia has never been purposely applied as a primary intervention in TBI patients.

This current study aims to assess the feasibility of conducting a single centre randomized controlled trial of TN versus no TN in traumatic brain injury (TBI) patients. Patients will be screened and enrolled through the trauma service in the Critical Care Trauma Centre (CCTC).

Patients who consent to enroll in the study will be randomized 1:1 into either the TN or no TN group. Participants allocated to the TN group will immediately commence targeted temperature management for 72 hours, with 4 hourly temperature checks and interventions as indicated. Participants in the no TN group will proceed with standard of care within CCTC. Both groups will be followed at 3 and 6 months post-discharge with cognitive assessments via the Creyos Health platform.

The trial will allow the research team to assess appropriate participant identification and enrollment rates, ease and limitations of intervention implementation, data collection, and post-discharge follow up. The research team will also assess the accessibility and ease of use of the Creyos Health platform in this patient population. In depth primary and secondary outcome measures are outlined elsewhere in the application.

This feasibility trial will be the first step in potentially introducing an evidence based intervention that directly targets cognitive outcomes in the TBI patient population group.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>= 18 years of age) who present through the LHSC trauma service and have sustained a TBI.
* A Glasgow Coma Scale (GCS) of 5-12, inclusive, prior to intubation.

Exclusion Criteria:

* GCS at time of presentation of 4 or less or 13 or more.
* Patients not expected to survive 48 hours.
* >24 hours from injury at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Study Execution | 18 months
  To assess the feasibility of conducting a randomized controlled trial of therapeutic normothermia compared to no therapeutic normothermia in LHSC patients with TBI.
Creyos Health | 12 months
  To assess the feasibility of using the Creyos Health platform as a cognitive assessment tool in patients with TBI.

SECONDARY OUTCOMES:
Mortality | 12 months.
  To assess any differences in in-hospital mortality between the two study groups.
Cognitive Outcomes | 12 months
  To assess any differences in cognitive outcomes between the two study groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ian Ball, MD, Principal Investigator — London Health Sciences Centre

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oshorov A, Baranich A, Polupan A, Sychev A, Savin I, Potapov A. Effects of Hyperthermia on Intracranial Pressure and Cerebral Autoregulation in Patients with an Acute Brain Injury. Acta Neurochir Suppl. 2021;131:71-74. doi: 10.1007/978-3-030-59436-7_15. PMID 33839821
- [Background] Hong JM, Choi ES, Park SY. Selective Brain Cooling: A New Horizon of Neuroprotection. Front Neurol. 2022 Jun 20;13:873165. doi: 10.3389/fneur.2022.873165. eCollection 2022. PMID 35795804
- [Background] Oshorov AV, Polupan AA, Sychev AA, Baranich AI, Kurdyumova NV, Abramov TA, Savin IA, Potapov AA. [Influence of cerebral hyperthermia on intracranial pressure and autoregulation of cerebral circulation in patients with acute brain injury]. Zh Vopr Neirokhir Im N N Burdenko. 2021;85(1):68-77. doi: 10.17116/neiro20218501168. Russian. PMID 33560622
- [Background] Nielsen N, Wetterslev J, Cronberg T, Erlinge D, Gasche Y, Hassager C, Horn J, Hovdenes J, Kjaergaard J, Kuiper M, Pellis T, Stammet P, Wanscher M, Wise MP, Aneman A, Al-Subaie N, Boesgaard S, Bro-Jeppesen J, Brunetti I, Bugge JF, Hingston CD, Juffermans NP, Koopmans M, Kober L, Langorgen J, Lilja G, Moller JE, Rundgren M, Rylander C, Smid O, Werer C, Winkel P, Friberg H; TTM Trial Investigators. Targeted temperature management at 33 degrees C versus 36 degrees C after cardiac arrest. N Engl J Med. 2013 Dec 5;369(23):2197-206. doi: 10.1056/NEJMoa1310519. Epub 2013 Nov 17. PMID 24237006
- [Background] Rosli D, Schnuriger B, Candinas D, Haltmeier T. The Impact of Accidental Hypothermia on Mortality in Trauma Patients Overall and Patients with Traumatic Brain Injury Specifically: A Systematic Review and Meta-Analysis. World J Surg. 2020 Dec;44(12):4106-4117. doi: 10.1007/s00268-020-05750-5. Epub 2020 Aug 28. PMID 32860141